CLINICAL TRIAL: NCT01681407
Title: Peripheral Plasma Micro-RNA and Proteomics Mapping in Depressive Patients, Treated With SSRI Medications.
Acronym: MIRPROT
Status: Terminated | Type: Observational
Why Stopped: Insufficient microRNA for the analysis
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amichai Hareven, Dr Amichai Hareven, HaEmek Medical Center, Israel
Other Study IDs: EMC-07411-CTIL
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Depression
Keywords: Depression; Selective Serotonin Reuptake Inhibitors; MicroRNAs; Proteome
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects and patients will be asked to give blood samples at 4 points of time for the lab processing: micro-RNA and proteome profiling/
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Depressed Patients: Patients: Group of patients that are diagnosed for having depression, and are suitable for SSRI treatment.
- Non-Depressed Controls: Controls: Volunteers that had clinical screening with no depression diagnosis.
- Patients Relatives: Patient Relatives (Optional group for later stage): First degree relatives with no depression diagnosis.

SUMMARY:
A pilot study of mapping the peripheral plasma micro-RNA and proteomics patterns in depressive patients, treated with SSRI medications. It is an observational clinical bio-markers laboratory controlled research with no device.

The research includes two groups; one for patients diagnosed of having depression, and will get a standard SSRI medication regimen. Second group is for control subjects without depression. An option for a third group is planned to include first degree relatives of the depressed patients. After giving their informed consents, subjects and patients will go through standard clinical psychiatric interview, and routine clinical lab tests. Clinical standard, specific depression and anxiety questionnaires will be held at four follow-up meetings: at start; after 2 weeks; 4 weeks; and 10 weeks. Subjects and patients will be asked to give blood samples at these points of time for the lab processing: Complete plasma proteomics and specific micro-RNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Depressed patients,over 18 yo
* Untreated with SSRI, in the last 3 months

Exclusion Criteria:

* Bipolar patients or another major psychopathology
* Depressive disorder clearly due to general medical condition, or drug related
* BMI under 18.5 or above 40
* Pregnant patients
* Active suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at community or hospital settings. Patients were clinically evaluated for suspected depression.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms remission or response rates, under usual SSRI treatment. | 10 weeks of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel